CLINICAL TRIAL: NCT03480178
Title: Renal Anemia Refractory to Erythropoietin
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, zaher alwi hadi, Assistant Lecturer, Assiut University
Other Study IDs: 17100366
Record Dates: First submitted 2018-02-13; First posted 2018-03-29 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: ESRD; Renal Anemia
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study evaluates the renal anemia refractory to Epo . in hemodialysis patients. all of participants will receive Epo. and identify various factors contributing to etiology of renal anemia in Epo- resistant patients.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is considered a public health problem worldwide with high incidence and prevalence rates.Anemia is one of the most frequent early complication of CKD. The main cause is erythropoietin (EPO) deficiency due to impaired kidney function However, other causes should be considered when the severity of anemia is inconsistent with the decrease in renal function; when there is evidence of iron deficiency or matching decreases in hemoglobin, leukopenia and/or thrombocytopenia are also found

ELIGIBILITY:
Inclusion Criteria:

* Patients greater than or equal to 18 years old with CKD on hemodialysis

Exclusion Criteria:

1. - Evidence of infections especial of vascular access .
2. - malnutrition and manifestation of iron, B12, folate and protein deficiency .
3. - any underling cause as;

   * Hematologic malignances -Hemolytic anemia -
   * Aplastic anemia (infection and/or bleeding with anemia)
   * Solid tumors
   * Bleeding (skin ,mucosal ,orificial)
   * Evidence of mineral bone disease (CKD-MBD)
   * Others

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. The investigators choose 50 uraemic patients on hemodialysis randomly and receiving Epo.among those admitted to nephrology ward and out Patient clinic of the department of internal medicine of Assiut University Hospital.
  2. Follow up of patients for 6 months with CBC every month.
  3. Searching for number of patients among this 50 who have failure to correct the anemia with Epo. (100IU /Kg / week- SC ) For target HB 11 gm.
  4. Effect of bleeding, infection and malnutrition.
  5. Scaring for the possible underling cause of anemia refractory to Epo. Clinically, laboratory at the end of study period.
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Renal anemia refractory to erythropoietin | 1 months
  1 .Measurement of Hemoglobin , feritin and reitculocyte of patient before treatmeant by Epo. 100IU per Kg per week-SC.
  2- Assessment to measure of hemoglobin of patient after treatment

SECONDARY OUTCOMES:
Renal anemia refractory to erythropoietin | 6MONTHS
  1 .Measurement of Hemoglobin of patient by CBC before treatmeant by Epo. 100IU per Kg per week-SC?
  2- Assessment to hemoglobin of anemic patient during the specified post -dose period ,6months

IPD SHARING:
Plan to Share IPD: No